CLINICAL TRIAL: NCT01588366
Title: Effects of LY2409021 on Hepatic Metabolism in Healthy Volunteers and Patients With Type 2 Diabetes Mellitus
Brief Title: The Effects of LY2409021 on the Liver
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13107; I1R-FW-GLBK (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — adomeglivant

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Part A and B - Up to 4 capsules of placebo administered orally once a day for 28 days.
  Interventions: Drug: Placebo
- 15 mg LY2409021 (Experimental): Part B - 1 capsule of 15 mg LY2409021 orally once a day for 28 days. (Arm added in September, 2012, per protocol amendment.)
  Interventions: Drug: LY2409021
- 60 mg LY2409021 (Experimental): Part A - 4 capsules of 15 mg LY2409021 administered orally once a day for 28 days.
  Interventions: Drug: LY2409021

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: LY2409021 — Administered orally
  Arms: 15 mg LY2409021; 60 mg LY2409021

SUMMARY:
This is a study that involves multiple doses of study drug (60 mg of LY2409021, 15 mg of LY2409021 or placebo) taken as capsules by mouth on a daily basis for 28 days. This study will image the liver using magnetic resonance imaging (MRI) and magnetic resonance spectroscopy (MRS) in healthy participants and in participants with type 2 diabetes mellitus, when they take LY2409021 to see if liver changes happen at the same time as changes in blood tests. This study is approximately 11 weeks long, not including screening. A screening appointment is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

For all participants:

* Must be a male, or a female who cannot become pregnant, and who is either a healthy participant, or who has type 2 diabetes
* Must have a body mass index (BMI) of 18.5 to 29.9 kilograms per square meter (kg/m^2) if a healthy participant, or a BMI of 18.5 to 35.0 kg/m^2 if diabetic

For participants with type 2 diabetes mellitus (T2DM):

- On diet and exercise treatment, or taking metformin

Exclusion Criteria:

For all participants:

* Have signs or symptoms of liver disease
* Are infected with hepatitis B or hepatitis C
* Have donated more than 450 mL of blood in the last 3 months or if have donated any blood in the last month
* Smoke more than 10 cigarettes per day or are not willing to abstain from smoking while at the clinic
* Have had surgery with metallic clips, staples or stents, or have had a cardiac pacemaker (or other surgical implants) inserted in any part of the body, or have fear of enclosed spaces or have symptoms that prevent them from being sent for an magnetic resonance imaging (MRI) scan

For participants with T2DM:

- Are using insulin

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started in April, 2012 with Part A. Part B was added per protocol amendment in September, 2012.
Groups:
- Placebo - Healthy (Part A): Placebo administered orally, once daily (QD) for 28 days to healthy participants.
- 60 mg LY2409021 - Healthy (Part A): 60 milligrams (mg) LY2409021 administered orally, QD for 28 days to healthy participants.
- Placebo - T2DM (Part A): Placebo administered orally, QD for 28 days to participants with type 2 diabetes mellitus (T2DM).
- 60 mg LY2409021 - T2DM (Part A): 60 mg LY2409021 administered orally, QD for 28 days to participants with T2DM.
- Placebo - T2DM (Part B): Placebo administered orally, QD for 28 days to participants with T2DM.
- 15 mg LY2409021 - T2DM (Part B): 15 mg LY2409021 administered orally, QD for 28 days to participants with T2DM.
Period: Overall Study
Arm/Group | Placebo - Healthy (Part A) | 60 mg LY2409021 - Healthy (Part A) | Placebo - T2DM (Part A) | 60 mg LY2409021 - T2DM (Part A) | Placebo - T2DM (Part B) | 15 mg LY2409021 - T2DM (Part B)
Started | 2 | 7 | 2 | 7 | 3 | 9
Received at Least One Dose of Study Drug | 2 | 7 | 2 | 7 | 3 | 9
Completed | 2 | 6 | 2 | 6 | 3 | 7
Not Completed | 0 | 1 | 0 | 1 | 0 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Placebo - Healthy (Part A): Placebo administered orally, QD for 28 days to healthy participants.
- 60 mg LY2409021 - Healthy (Part A): 60 mg LY2409021 administered orally, QD for 28 days to healthy participants.
- Placebo - T2DM (Parts A and B): Placebo administered orally, QD for 28 days to participants with T2DM.
- Total: Total of all reporting groups
Arm/Group | Placebo - Healthy (Part A) | 60 mg LY2409021 - Healthy (Part A) | Placebo - T2DM (Parts A and B) | 15 mg LY2409021 - T2DM (Part B) | 60 mg LY2409021 - T2DM (Part A) | Total
Number analyzed (Participants) | 2 | 7 | 5 | 9 | 7 | 30
Age, Continuous [Mean (Standard Deviation); unit: years]
  Healthy Participants | 49.5 (13.4) | 39.3 (13.2) | NA (NA) — Row represents healthy participants only | NA (NA) — Row represents healthy participants only | NA (NA) — Row represents healthy participants only | 41.6 (13.2)
  T2DM subjects | NA (NA) — Row represents T2DM subjects only | NA (NA) — Row represents T2DM subjects only | 60.0 (5.1) | 55.7 (7.9) | 51.4 (10.0) | 55.3 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 1 | 2 | 4
  Male | 2 | 7 | 4 | 8 | 5 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 5 | 9 | 7 | 30
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 2 | 7 | 5 | 9 | 7 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 28 in Liver Fat Average Percent (%)
Description: Measured by magnetic resonance (MR) scanning.
Time Frame: Baseline, Day 28 (Pre-meal)
Population: All participants who had evaluable MR scans at Baseline and on Day 28.
Measure: Mean (95% Confidence Interval); unit: percentage of liver fat average
Arm/Group | Placebo - Healthy (Part A) | 60 mg LY2409021 - Healthy (Part A) | Placebo - T2DM (Parts A and B) | 15 mg LY2409021 - T2DM (Part B) | 60 mg LY2409021 - T2DM (Part A)
Number analyzed (Participants) | 2 | 6 | 5 | 7 | 6
percentage of liver fat average | -0.47 [NA to NA] — For n=2, confidence Intervals were not calculated due to few participants. | 5.55 [0.346 to 10.7] | -1.49 [-5.00 to 2.03] | 4.45 [1.66 to 7.24] | 5.84 [3.17 to 8.51]

2. Primary Outcome: Change From Baseline to Day 28 in Hepatic Glycogen Content
Description: Measured by MR scanning.
Time Frame: Baseline, Day 28 (Pre-meal)
Population: All participants in Part A who received 60 mg LY2409021 and had evaluable MR scans at Baseline and on Day 28.
Measure: Mean (95% Confidence Interval); unit: millimoles per liter (mmol/L)
Arm/Group | 60 mg LY2409021 - Healthy (Part A) | 60 mg LY2409021 - T2DM (Part A)
Number analyzed (Participants) | 6 | 5
millimoles per liter (mmol/L) | 12.8 [-48.1 to 73.8] | 42.1 [-8.18 to 92.4]

3. Secondary Outcome: Change From Baseline to Day 28 in Transaminase Levels
Time Frame: Baseline, Day 28
Population: All participants who had evaluable transaminase levels at Baseline and on Day 28.
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | Placebo - Healthy (Part A) | 60 mg LY2409021 - Healthy (Part A) | Placebo - T2DM (Parts A and B) | 15 mg LY2409021 - T2DM (Part B) | 60 mg LY2409021 - T2DM (Part A)
Number analyzed (Participants) | 2 | 6 | 5 | 7 | 6
units per liter (U/L)
  Alanine aminotransferase (ALT) | -0.5 (0.7) | 47.7 (51.6) | -3.5 (4.3) | 15.7 (15.1) | 13.3 (5.8)
  Aspartate aminotransferase (AST) | 0.3 (3.2) | 22.2 (22.8) | -0.2 (3.7) | 9.9 (9.5) | 7.7 (4.8)

4. Secondary Outcome: Change From Baseline to Day 29 in Glucose Response to an Arginine Stimulation Test (AST) (Part A)
Description: Acute glucose response to an AST at a blood glucose level of approximately 250 milligrams per deciliter (mg/dL).
Time Frame: Baseline, Day 29
Population: Zero participants were analyzed for this outcome measure because glucose response data was not collected or included in the data analysis plan.
Groups:
- 60 mg LY2409021 (Healthy): Part A: 60 mg LY2409021 administered orally, QD, for 28 days in healthy participants.
- 60 mg LY2409021 (T2DM): Part B: 60 mg LY2409021 administered orally, QD for 28 days in participants with T2DM.
Arm/Group | 60 mg LY2409021 (Healthy) | 60 mg LY2409021 (T2DM)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline to Day 29 in Glucagon Response to an Arginine Stimulation Test (AST) (Part A)
Description: Acute glucagon response to an AST at a blood glucose level of approximately 250 mg/dL.
Time Frame: Baseline, Day 29
Population: All participants in Part A who received 60 mg LY2409021 and had an evaluable glucagon response at Baseline and on Day 29.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | 60 mg LY2409021 - Healthy (Part A) | 60 mg LY2409021 - T2DM (Part A)
Number analyzed (Participants) | 5 | 7
pmol/L | 80.0 [42.2 to 118] | 103 [79.5 to 126]

6. Secondary Outcome: Change From Baseline to Day 29 in Insulin Response to an Arginine Stimulation Test (AST) (Part A)
Description: Acute insulin response to an AST at a blood glucose level of approximately 250 mg/dL.
Time Frame: Baseline, Day 29
Population: All participants in Part A who received 60 mg LY2409021 and had an evaluable insulin response at Baseline and on Day 29.
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | 60 mg LY2409021 - Healthy (Part A) | 60 mg LY2409021 - T2DM (Part A)
Number analyzed (Participants) | 5 | 7
pmol/L | -34.7 [-207 to 138] | 139 [-73.6 to 352]

ADVERSE EVENTS:
Arm/Group | Placebo - Healthy (Part A) | 60 mg LY2409021 - Healthy (Part A) | Placebo - T2DM (Parts A and B) | 15 mg LY2409021 - T2DM (Part B) | 60 mg LY2409021 - T2DM (Part A)
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/7 | 0/5 | 2/9 | 0/7
Other Adverse Events (participants affected / at risk) | 1/2 | 7/7 | 4/5 | 7/9 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Healthy (Part A) (N=2) | 60 mg LY2409021 - Healthy (Part A) (N=7) | Placebo - T2DM (Parts A and B) (N=5) | 15 mg LY2409021 - T2DM (Part B) (N=9) | 60 mg LY2409021 - T2DM (Part A) (N=7)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Healthy (Part A) (N=2) | 60 mg LY2409021 - Healthy (Part A) (N=7) | Placebo - T2DM (Parts A and B) (N=5) | 15 mg LY2409021 - T2DM (Part B) (N=9) | 60 mg LY2409021 - T2DM (Part A) (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 2 (3)
Catheter site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Vessel puncture site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes